CLINICAL TRIAL: NCT04180553
Title: Ultrasound-Guided Resuscitation in Open Aortic Surgery
Acronym: AORTUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Luc Dubois, Principal Investigator, London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 113875
Record Dates: First submitted 2019-10-22; First posted 2019-11-27 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Aortic Diseases
Keywords: Ultrasound; Goal-directed resuscitation
MeSH Terms: conditions — Aortic Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial - 20 patients per arm. A permuted block randomization plan will be used with block sizes of 2 and 4
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Point-Of-Care Ultrasound Guided Resuscitation (Experimental): Intervention in this trial is randomization to POCUS management for goal-directed post-operative resuscitation for the first 48 hours of admission.Patients randomized to the use of POCUS will have a focused cardiac, thoracic, and IVC study performed post-operatively in PACU, as well as regular (BID) assessments on the inpatient ward for post-operative day one and two. Based on ultrasound findings, their fluid resuscitation will be guided to a fluid liberal or fluid restrictive strategy at the time of each assessment.
  Interventions: Diagnostic Test: Point of Care Ultrasound (POCUS)
- Usual Care (Active Comparator): The comparator arm in this trial is randomization to usual care. Participants randomized to control group for usual care will undergo resuscitation guided by modalities used currently, which can include both static and dynamic measures. These will include review of vital signs, biochemistry, and urine output as well as bedside physical exam. In this arm, patients will not undergo POCUS during their admission. IV fluid infusion rates as well as targets for IV boluses will be left to the discretion of the attending physician and can include hypotension, hypovolemia, as well as oliguria
  Interventions: Other: Usual Care

INTERVENTIONS:
Diagnostic Test: Point of Care Ultrasound (POCUS) — The intervention group will receive a 4-view transthoracic echocardiogram including Parasternal long axis, parasternal short axis, apical 4-chamber, and supplemental subcostal short-axis/4-chamber views as needed. A standard 4-view thoracic lung ultrasound study will assess the left and right anterior chest wall, anterior axillary regions, as well as the costophrenic angle and posterolateral regions. At 5 discrete time intervals post-operatively, POCUS assessments will be used to adjust fluid resuscitation to fluid liberal (2cc/kg/hr) or fluid restrictive (0.8cc/kg/hr). Routine vital signs, biochemistry, and urine output as well as bedside physical exam will be assessed as usual. IV boluses of crystalloid will be permitted to treat hypotension with SBP <90mmHg with clinical signs of hypovolemia, but oliguria will not be used as a marker to titrate fluid infusion rates. Blood transfusion may be used for post-operative bleeding or anemia as clinically indicated.
  Arms: Point-Of-Care Ultrasound Guided Resuscitation
Other: Usual Care — The control group for "usual care" will undergo resuscitation guided by modalities used currently, which can include both static and dynamic measures. These will include review of vital signs, biochemistry, and urine output as well as bedside physical exam. In this arm, patients will not undergo POCUS during their admission. IV fluid infusion rates as well as targets for IV boluses will be left to the discretion of the attending physician and can include hypotension, hypovolemia, as well as oliguria. Blood transfusion may be used for post-operative bleeding or anemia as clinically indicated.
  Arms: Usual Care

SUMMARY:
This study will aim to determine whether routine Point of Care Ultrasound (POCUS) assessment of volume status, cardiac function, and pulmonary function after major abdominal aortic surgery is an accurate and feasible form of monitoring for individualized, goal-directed resuscitation. Half of the patients will receive POCUS-guided fluid resuscitation, and the other half will be resuscitated using usual post-operative care.

DETAILED DESCRIPTION:
Patients assessed for elective open aortic surgery for both aneurysmal and occlusive disease either as inpatients or in the outpatient vascular surgery clinic will be screened for eligibility at the time of initial consultation. Once the patient has been screened for eligibility, the participant will be enrolled on the basis of informed consent with a letter of information. This study will be submitted for review by the Health Sciences Research Ethics Board at Western University. This will be a feasibility trial, with the primary endpoints reflecting safety and feasibility outcomes of executing the trial protocol as outlined in this document.

Intervention in this trial is randomization to POCUS management for goal-directed post-operative resuscitation for the first 48 hours of admission, whereas the control group will be management by usual care for the first 48 hours of admission. Patients randomized to the use of POCUS will have a focused cardiac, thoracic, and Inferior vena cava (IVC) study performed post-operatively in the surgery recovery room, as well as regular (BID) assessments on the inpatient ward for post-operative day one and two.

The protocol for the intervention group will receive a 4-view transthoracic echocardiogram including the following views: Parasternal long axis, parasternal short axis, apical 4-chamber, and supplemental subcostal short-axis and subcostal 4-chamber if parasternal views are limited. Color Doppler will be used for qualitative valvular assessment if indicated. A longitudinal IVC view will be obtained in the usual subcostal transabdominal position, or the transhepatic position if the transabdominal view is not technically feasible. A thoracic lung ultrasound study will assess the left and right anterior chest wall, anterior axillary regions, as well as the costophrenic angle and posterolateral regions. Participants randomized to the point of care ultrasound arm will also have access to routine avenues of patient assessment which include review of vital signs, biochemistry, and urine output as well as bedside physical exam. Images acquired will be overread by sonographic experts with expertise in bedside point of care echocardiography through a central image reporting system.

Point of care studies will synthesize cardiac, thoracic, and IVC views to elucidate whether patients who fluid deplete or fluid replete, and if ventricular dysfunction is contributing to hypotension or end-organ dysfunction. They will be allocated to either a fluid restrictive or fluid liberal management strategy accordingly. The fluid liberal group will receive a fluid infusion of 2ml/kg/hr of balanced crystalloid solution. For patients with a body weight greater than 100kg, fluid volumes will be calculated based on a maximum body weight of 100kg. The fluid restrictive group will receive a fluid infusion of 0.8ml/kg/hr of balanced crystalloid solution. IV boluses of crystalloid will be permitted to treat hypotension with systolic blood pressure <90 with clinical signs of hypovolemia, but oliguria will not be used as a marker to titrate fluid infusion rates. Blood transfusions will be permitted to treat post-operative bleeding or anemia as clinically indicated. Those with severely decreased left ventricular function who are presumed to be hypotensive secondary to poor cardiac output will be transferred to an appropriate level 1 care monitored bed to receive vasopressors or inotropes to manage their hypotension. They will be managed to the fluid restrictive arm with an infusion rate of 0.8 ml/kg/hr of ringer's lactate solution. Once all patients are able to tolerate oral fluid intake, their maintenance IV fluid infusions will be discontinued.

Participants randomized to control group for usual care will undergo resuscitation guided by modalities used currently, which can include both static and dynamic measures. These will include review of vital signs, biochemistry, and urine output as well as bedside physical exam. In this arm, patients will not undergo POCUS during their admission. IV fluid infusion rates as well as targets for IV boluses will be left to the discretion of the attending physician and can include hypotension, hypovolemia, as well as oliguria. Blood transfusion may be used for post-operative bleeding or anemia as clinically indicated.

This protocol does not restrict formal radiographic or ultrasound studies such as plain film x-rays, CT, MRI, echocardiography, abdominal ultrasonography, and duplex ultrasound of lower extremity veins in patients in the intervention or control groups with appropriate clinical indications.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older.

  o There is no upper age limit for eligibility in this study.
* Elective surgical procedures
* Patients who are enrolled must be receiving open abdominal surgery for either occlusive disease (aortobifemoral bypass, transaortic endarterectomy) or aneurysmal disease (infrarenal, juxtarenal abdominal aortic aneurysms).
* Patients must be deemed suitable operative candidates for open abdominal aortic surgery as decided upon by the surgical and perioperative medicine assessments.

Exclusion Criteria:

* Thoracoabdominal aneurysms (Type IV or larger extent)
* Hybrid procedures (Requiring both endovascular and open surgical reconstruction)
* Pediatric vascular cases (Patients less than 18 years of age)
* Emergency cases
* American Society of Anesthesia (ASA) class 5 identified
* Chronic renal failure requiring dialysis
* Inability of patient to consent to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Recruitment | 30 days
  Recruitment - Overall proportion of eligible patients successfully entered into the study divided by the total number of eligible patients consented and retained to full data completion - ≥80% recruitment rate
Feasibility - Successful Randomization | 30 days
  Overall proportion of consented patients successfully receiving randomization at the completion of operation divided by the total number of consented patients - ≥80% randomized
Feasibility - POCUS Study completion | 30 days
  Overall proportion of completed studies divided by expected studies - ≥80% completion
Feasibility - Protocol Adherence | 30 days
  Overall proportion of patients adequately receiving treatment as defined by the trial protocol divided by the total number of patients enrolled - ≥80% Adherence
Feasibility - Successful Data Collection | 30 days
  Overall proportion of patients with no absent data points in the database divided by the total number of patients enrolled - ≥80% complete data sets
Feasibility - Contamination rate | 30 days
  The number of patients crossed over into the opposite arm of the study based on patient or physician motivators divided by the total number of patients enrolled - ≤20% contamination

SECONDARY OUTCOMES:
Feasibility - POCUS image quality | 30 days
  Image quality - Agreement between physicians performing POCUS and experts auditing studies will be measured for both image acquisition and interpretation - ≥80% agreement

CONTACTS AND LOCATIONS:
Overall Officials: Luc Dubois, MD, Principal Investigator — London Health Sciences Center
Locations (1):
- London Health Sciences Center - Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
As this is a feasibility trial, there are no plans to make individual patient data available to other researchers. The individual patient data may be used as part of a larger randomized controlled trial if the feasibility trial shows the protocol is feasible and safe.